CLINICAL TRIAL: NCT01671345
Title: A Randomized Trial of an Educational Intervention in Type 2 Diabetes Patients
Brief Title: An Educational Intervention for Type 2 Diabetes Patients
Acronym: ACTIVet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IIR 12-050
Record Dates: First submitted 2012-06-14; First posted 2012-08-23 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Patients randomized to the intervention will view the intervention video
  Interventions: Behavioral: Intervention Video
- Control (Placebo Comparator): Patients randomized to control will view an informative video about nutrition and exercise of similar length
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention Video — A video intervention delivered prior to patients' visits with primary care physicians designed to increase use of active participatory communication (patient participation) behaviors, improved communication ratings, and improved medication adherence
  Other Names: Speak Up!
  Arms: Intervention
Behavioral: Control — Attention control
  Arms: Control

SUMMARY:
Diabetes is common, it is expensive, and it is a chronic condition. Estimates put the prevalence of diabetes at almost 20 percent in VA patients and the prevalence of diabetes in the VA is higher among racial and ethnic minorities. Poorly controlled diabetes leads to a number of complications including cardiovascular disease, blindness, amputation, and end stage renal disease. Adherence to medication regimens (as well as lifestyle factors such as diet and exercise) is important to achieve diabetes care goals. Adherence to recommended care is related at least in part to effective communication in medical encounters. This project is designed to test a video intervention to improve patients' communication behaviors. Doctors will also receive a communication skills training program. The project will assess the impact of the training programs on communication and outcomes. The study is designed to help make patient care more patient-centered, which is one of the six aims for improvement in the Institute Of Medicine report, Crossing the Quality Chasm and is a goal of VA transformation efforts.

DETAILED DESCRIPTION:
Background: Diabetes is estimated to affect up to 1 in 5 VA patients overall and up to 1 in 4 racial/ethnic minority patients. Patients with low health literacy and minority groups have more difficulty communicating with physicians, report lower adherence to physicians' recommendations, and have higher rates of poor diabetes outcomes. Activating patients to use more effective communication with physicians' can lead to better adherence to treatment and to better biomedical outcomes. In this project the investigators build upon their prior work from two Health Services Research & Development (HSRD) funded pilot projects to improve doctor patient communication in patients with type 2 diabetes mellitus (T2DM). In a previously funded short-term project, #SHP-08-182, the investigators conducted focus groups with patients with T2DM to elicit and understand from the patient perspective, barriers to communicating with their physician. This qualitative work was used in a subsequent pilot project, #PPO-08-402 to refine and pilot test an educational video to encourage patients to use active participatory communication in their visits to physicians. This work was successfully completed and the product is a 10 minute video that in testing was found to be acceptable to patients and feasible for patients to view immediately preceding their medical encounter.

Objectives: In this project the investigators propose to test the effectiveness of the video as an intervention to improved patients' communication. The primary aim is to conduct a randomized controlled trial of an intervention testing whether the intervention increases patients' active participatory communication behaviors, patients' post-visit ratings of self efficacy to communicate, medication adherence, and diabetic control (HgbA1c). There are four secondary aims which include assessments of the (1) mediators, and (2) moderators of the relationship of the intervention condition to outcomes, (3) costs of the intervention, and (4) an evaluation of the feasibility of using the video for pre-visit preparation.

Methods: The investigators will conduct a two group, pre-post, randomized controlled, single-site trial of the intervention in patients with T2DM. The investigators will recruit 156 patients and their physicians for a pre and post-intervention visit. Physicians will be trained with the agenda setting module from the Four Habits model. Patients will be randomized to view a 10 minute intervention or control video prior to their second visit. Visits will be audio recorded and analyzed for patients' and physicians' communication behaviors. Self-efficacy to communicate will be collected by self report. Adherence will be collected by self-report and by medication possession ratio. Diabetic control is collected by chart review. Analyses will evaluate the relationship of the intervention condition to outcomes, mediators and moderators of that relationship, and will estimate costs of the intervention and feasibility of using the video in a busy clinic.

Impacts: VA transformation efforts including interprofessional Patient Aligned Care Teams (PACT) are focusing attention on patient-centered care. Improved communication is a central feature of patient centered care. Communication in medical interactions is critical and plays an important, but often overlooked role in health-care decision making and quality of care. Patients who have difficulty communicating are less involved in consultations with their physician, receive less information and support, and are less satisfied with their care. In turn, these patients may not understand their treatment options, may have less knowledge, less positive beliefs about treatment and less trust in physician, and may experience poorer health outcomes. Teaching patients to communicate more effectively is patient-centered because it inherently supports a patient-driven approach to delivering healthcare. The investigators' intervention is designed to encourage patients' active communication. Improving patients' communication is a unique focus that may supplement and add to the VA efforts in areas such as the Patient Aligned Care Team. In addition, the methodology is not disease specific and may be a paradigm for improvement in other conditions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* Hemoglobin A1c (HgbA1c) greater than or equal to 8
* Adults, age 18 or older

Exclusion Criteria:

* Lives in skilled nursing facility
* Dementia (abnormal score on Mini-COG)
* Terminal medical condition
* Drug- (e.g., steroid) induced diabetes.
* Blind or deaf (e.g., unable to view/hear video)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2013-11-27 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Gordon, MD SB, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gordon HS, Street RL. How Physicians, Patients, and Observers Compare on the Use of Qualitative and Quantitative Measures of Physician-Patient Communication. Eval Health Prof. 2016 Dec;39(4):496-511. doi: 10.1177/0163278715625737. Epub 2016 Jan 10. PMID 26755527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients (active diagnosis of type 2 diabetes mellitus and a hemoglobin A1c ≥ 7.5) were identified and recruited from the Primary Care clinic and Women's clinics at the Jesse Brown Veterans Affairs Medical Center (JBVAMC) in Chicago. Recruitment period lasted from 11/27/13 to 11/30/16.
Pre-assignment Details: 794 patients were screened; 625 were excluded (not meeting inclusion criteria -188, declined participation/did not respond to invite - 437). 169 patients were enrolled.
Groups:
- Intervention: Patients randomized to the intervention view the intervention video.
  Intervention Video: A video intervention delivered prior to patients' visits with primary care physicians designed to increase use of active participatory communication (patient participation) behaviors, improved communication ratings, and improved medication adherence.
- Control: Patients randomized to control view an informative video about diet and nutrition of similar length.
  Control: Attention control.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 77 | 92
Completed | 64 | 83
Not Completed | 13 | 9
Not completed — Lost to Follow-up | 10 | 6
Not completed — visit with non-participating physician | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 64 | 83 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 57 | 100
  >=65 years | 21 | 26 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.19 (7.78) | 59.50 (8.21) | 59.89 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 54 | 71 | 125
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 64 | 83 | 147

OUTCOME MEASURES:

1. Primary Outcome: Patients' Perceived Self-efficacy to Communicate
Description: Communication Self-Efficacy is the degree to which a patient feels able to interact with his/her physician in order to provide information about problems, obtain desired information about diagnosis, treatment and prognosis, and participate in formulating a plan. Self Efficacy to Communicate is measured with the Perceived Efficacy in Physician Patient Interactions scale - a valid and reliable self report measure of patients' perceived self efficacy in interacting with physicians. Scores ranging from 5 to 25 are used; higher numbers reflect more perceived self-efficacy in interacting with physicians.
Time Frame: at the baseline ( Visit 1) and post-intervention (Visit 2)
Population: Patients with type 2 diabetes and with HgbA1c more than or equal to 7.5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 64 | 83
units on a scale
  Visit 1 | 22.11 (3.24) | 22.14 (3.06)
  Visit 2 | 23.44 (2.40) | 22.63 (2.99)

2. Primary Outcome: Patients Active Participatory Communication Behaviors
Description: Active Participatory Communication Behavior (collected at visits 1 and 2) is derived from the content of audio recordings of the physician-patient visits.
  Active participatory communication behaviors include four essential elements:
  1. telling a medical history;
  2. asking questions;
  3. being assertive or making requests, and
  4. communication concerns. We coded patients' active participatory communication behaviors from the audio recording by classifying patients' statements into utterances. An utterance is the unit of analysis for coding the different types of behaviors into the communication categories. Utterances are coded according to the categories of active participatory communication behavior. Once classified, communicative behaviors are summed. The higher number means more active communication.
Time Frame: at the baseline ( Visit 1) and post-intervention (Visit 2)
Population: Patients with type 2 diabetes at JBVAMC with HgbA1c more than or equal 7.5
Measure: Mean (Standard Deviation); unit: utterances
Arm/Group | Intervention | Control
Number analyzed (Participants) | 64 | 83
utterances
  Visit 1 | 41.96 (25.89) | 44.32 (29.25)
  Visit 2 | 43.02 (30.95) | 42.92 (26.52)

3. Secondary Outcome: Medication Adherence
Description: Patient adherence to medication was measured with: (1) Medical Outcome Study measure and (2) Morisky scale.
  1. The Medical Outcome Study self-reported adherence to physicians' recommendations scale uses a brief questionnaire that asks whether respondents were adherent to physicians' recommendations and has scores ranging from 25 to 100. Higher numbers reflect better adherence.
  2. The Morisky scale (4-item version) assesses self-reported medication adherence using "yes" or "no" questions to evaluate how a patient feels when they stop taking medication, if they feel hassled about taking medication, and if they have difficulty remembering to take their medication. The scores range form 0 to 4; higher numbers reflect better adherence.
Time Frame: Four weeks post-intervention (i.e. four weeks after Visit 2).
Population: Patients with type 2 diabetes at JBVAMC with HgbA1c more than or equal to 7.5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention: Patients randomized to the intervention view the intervention video
  Intervention Video: A video intervention delivered prior to patients' visit 2 with primary care physician designed to increase use of active participatory communication (patient participation) behaviors, improved communication ratings, and improved medication adherence
Arm/Group | Intervention | Control
Number analyzed (Participants) | 64 | 83
units on a scale
  Measure of Outcome study: number analyzed (Participants) | 64 | 82
  Measure of Outcome study | 82.66 (14.31) | 78.78 (18.80)
  Morisky scale: number analyzed (Participants) | 64 | 82
  Morisky scale | 3.26 (1.03) | 3.23 (0.92)

4. Secondary Outcome: Hemoglobin A1c
Description: Hemoglobin A1c (HgbA1c) is the blood test for assessing the control of diabetes over approximately three months preceding the test. HgbA1c is usually checked many times a year in patients with poorly controlled diabetes. Baseline HgbA1c in patients had to be ≥ 7.5.
Time Frame: At the baseline (Visit 1) and post-intervention (after Visit 2). All available values were restricted to one year before Visit 1 and from 30 days to one year past Visit 2.
Population: Patients with type 2 diabetes at JBVAMC with HgbA1c more than or equal 7.5
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Intervention: Patients randomized to the intervention view the intervention video
  Intervention Video: A video intervention delivered prior to patients' visits with primary care physicians designed to increase use of active participatory communication (patient participation) behaviors, improved communication ratings, and improved medication adherence.
- Control: Patients randomized to control view an informative video about diet and nutrition of similar length
  Control: Attention control
Arm/Group | Intervention | Control
Number analyzed (Participants) | 64 | 83
percent
  baseline | 10.07 (1.93) | 9.53 (1.31)
  post-visit 2 | 9.07 (1.68) | 9.27 (1.73)

ADVERSE EVENTS:
Time Frame: From the baseline (Visit 1) to the follow-up telephone interview that was conducted four weeks post-intervention (i.e. four weeks after Visit 2). As this is a pragmatic study, we could not enforce the same specific time interval on each patient. Time frame varies depending on occurrence of patients' appointments with their physicians in routine clinical practice.
Groups:
- Control: Patients randomized to control will view an informative video about diet and nutrition of similar length.
  Control: Attention control.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/92
Other Adverse Events (participants affected / at risk) | 0/77 | 0/92

LIMITATIONS AND CAVEATS:
The analysis of communication outcomes is not yet complete because of delays in coding of transcribed audio-recordings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes